CLINICAL TRIAL: NCT06757907
Title: Topical Ganciclovir Versus Systemic Aciclovir in the Treatment of Herpetic Keratitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab Tharwat, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Herpetic Keratitis
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Herpetic Keratitis
Keywords: acyclovir; ganciclovir
MeSH Terms: conditions — Keratitis, Herpetic; Multiple Acyl Coenzyme A Dehydrogenase Deficiency | interventions — Acyclovir; Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ganciclovir (Active Comparator)
  Interventions: Drug: Ganciclovir (GCV)
- Systemic acyclovir (Active Comparator)
  Interventions: Drug: Acyclovir 400 MG

INTERVENTIONS:
Drug: Acyclovir 400 MG — Acyclovir is used to treat infections caused by certain types of viruses.
  Arms: Systemic acyclovir
Drug: Ganciclovir (GCV) — Ganciclovir is an anti-viral drug
  Arms: ganciclovir

SUMMARY:
Traditional antiviral treatments, including systemic acyclovir, have shown effectiveness in resolving keratitis but can also lead to complications, including ocular surface toxicity and the development of acyclovir-resistant strains of HSV. Topical ganciclovir 0.15% ophthalmic gel presents a safer alternative for managing herpetic keratitis, offering effective viral suppression with minimal toxicity. This study aims to compare the efficacy and safety of topical ganciclovir versus systemic acyclovir in treating herpetic keratitis, providing valuable insights into optimal management strategies for this condition

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with herpetic keratitis

Exclusion Criteria:

* Patients with known allergies to ganciclovir or acyclovir
* Severe ocular surface disease
* Those who have previously received antiviral therapy for herpetic keratitis within the last month

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Corneal healing | At 4 and 6 weeks
  Heling of the keratitis

SECONDARY OUTCOMES:
Sie effects | at 4 and 6 weeks
  Measuring the percentage of the side effects of the drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar university, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided